CLINICAL TRIAL: NCT06575517
Title: A Multifaceted Intervention to Improve Bleeding Management Among Patients Using Oral Anticoagulants (IMPACT-BLEEDING): a Cluster-randomized Trial
Brief Title: A Multifaceted Intervention to Improve Bleeding Management Among Patients Using Oral Anticoagulants (IMPACT-BLEEDING)
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn due to a realignment of strategic priorities.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9603R00021
Record Dates: First submitted 2024-08-01; First posted 2024-08-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The Group 1 in this trial will consist of a multifaceted bundle of instructions to sites about optimal management of bleeding.
- Group 2: The Group 2 will be randomized to the standard of care. Standard of care will be left to the discretion of the sites (clusters) participating in the study.

SUMMARY:
Prospective, cluster randomized trial including expected 168 patients with chronic use of oral anticoagulation (OAC) suffering major bleeding. Randomization will be performed stratified by geographic region (Southern/Southeastern Brazil versus other Brazilian regions).

DETAILED DESCRIPTION:
The Group 1 in this trial will consist of a multifaceted bundle of instructions to sites about optimal management of bleeding, including transfusion thresholds and when indicated; laboratory assessment of coagulation when indicated; reversal agents when indicated, and tailored approach to restarting of oral anticoagulation and dosing adjustments among patients after bleeding episode. This bundle will be based on a society guideline on bleeding management from the American College of Cardiology. The Group 2 will be randomized to the standard of care. Standard of care will be left to the discretion of the sites (clusters) participating in the study. All sites, including those from the control group, will be encouraged to follow local policies of blood product utilization and bleeding management.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years;
* Patients using chronic OAC (that is, for 30 or more consecutive days) due to AF/flutter, VTE or other clinical indication and presenting with a major bleeding episode according to the definition of the International Society of Thrombosis and Hemostasis (ISTH). Exclusion criteria
* Patients with limitation to follow-up;
* Patients with do not resuscitate order at time of enrolment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic use of oral anticoagulant (OAC) suffering a major bleeding event while on OAC.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients adherent to a predefined checklist for optimal bleeding management strategies | 2 months
  This checklist will involve proper use of blood products; proper use of reversal agents; proper dose adjusting and timing of restart of anticoagulation.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home